CLINICAL TRIAL: NCT05574231
Title: A Danish Nationwide Longitudinal Registered Based Study on Prevalence, Treatment Patterns and Disease Trajectories of Periodontitis and Co-morbidities 'PlanPerioMed'
Brief Title: A Danish Nationwide Longitudinal Study on Prevalence of Periodontitis and Its Co-morbidities
Acronym: PlanPerioMed
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: Plandent A/S (Unknown)
Responsible Party: Principal Investigator, Christian Damgaard, Associate professor, Head of Section, University of Copenhagen
Other Study IDs: 522-0018/22-3800; 522-0018/22-3800 (Other Grant/Funding Number: Plandent A/S)
Record Dates: First submitted 2022-09-01; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Periodontitis; Diabetes Mellitus, Type 2; Cardiovascular Diseases; Rheumatoid Arthritis
Keywords: Periodontal Diseases, Periodontal Index, Periodontal Bone Loss, Periodontal Attachment Loss, Probing Depth, Bleeding on Probing, Clinical Attachment Loss; Diabetes Mellitus 2, DM type 2, Non-insulin dependent diabetes mellitus, Uncontrolled diabetes mellitus type 2, Increased blood glucose level; CVD, Cardiovascular risk, Heart disease, Heart disease risk factors; Smoking status, Socio-economic status, Register based, Longitudinal study, Danish nationwide study, systemic diseases
MeSH Terms: conditions — Periodontitis; Diabetes Mellitus, Type 2; Cardiovascular Diseases; Arthritis, Rheumatoid; Periodontal Diseases; Alveolar Bone Loss; Periodontal Attachment Loss; Heart Diseases | interventions — Periodontal Index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 25 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Periodontal treatment — It includes surgical and non-surgical procedures depending on patient as well as tooth level.

SUMMARY:
The project (PlanPerioMed) is a register-based study evaluating the associations and patterns of health care delivery between periodontitis and medical diseases using data from the Danish dental record system Dentalsuite (Plandent A/S) and national Danish health care registries with three overall hypotheses/ aims:

* Determine the extent to which periodontitis in registry data is associated with more odontological treatment services and treatment frequency.
* Determine if patients with systemic diseases attend dentists more frequently and receive more treatment services per patient than the population without these diseases.
* Determine to which extent periodontitis and received periodontal treatment affects the risk of medical diseases.

The study will focus on association and trajectories of periodontitis and its treatment with three medical diseases, namely, Type 2 Diabetes Mellitus (Type 2 DM), Cardiovascular Diseases (CVD) and Rheumatoid Arthritis (RA). The dataset consists of approximately 4,000,000 people aged between 18 and 99 years attending private practice in Denmark. The results from PlanPerioMed study are likely to have ramifications for treatment guidelines for other periodontitis comorbidities, e.g. CVD and DM, and will thereby improve the quality of life for a wide range of patients and reduce long-term societal health care expenses related to periodontitis and its comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with clinical registrations of DMFT, periodontal status and corresponding treatment codes
* Self-reported systemic diseases including Diabetes Mellitus Type 2, Cardiovascular Diseases and Rheumatoid Arthritis
* Subjects with Clinical Attachment Loss>=3mm, Probing Depth >= 3mm and bleeding on probing (as defined by World Workshop 2017- criteria for periodontitis) in clinical examination will be included in the study population.

Exclusion Criteria:

* Subjects with more than 32 teeth
* Subjects with no clinical registrations

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include people who are clinically diagnosed with periodontal diseases and private practice dental care attenders in Denmark.
Sampling Method: Probability Sample
Enrollment: 4000000 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment frequency and type of treatment services | 25 years
  Number of treatment and odontological treatment services due to periodontitis
Treatment frequency and type of treatment services among patients with medical diseases | 25 years
  Number of treatment and odontological treatment services among patients with medical diseases due to periodontitis
Effect on medical diseases | 25 years
  Risk of medical diseases based on periodontal disease extent and received periodontal treatment

CONTACTS AND LOCATIONS:
Overall Officials: Anne Havemose Poulsen, Study Director — Head of Department

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kongstad J, Ekstrand K, Qvist V, Christensen LB, Cortsen B, Gronbaek M, Holm-Pedersen P, Holmstrup P, Bardow A, Twetman S, Fiehn NE. Findings from the oral health study of the Danish Health Examination Survey 2007-2008. Acta Odontol Scand. 2013 Nov;71(6):1560-9. doi: 10.3109/00016357.2013.776701. Epub 2013 Apr 29. PMID 23627881
- [Background] Kongstad J, Enevold C, Christensen LB, Fiehn NE, Holmstrup P. Impact of Periodontitis Case Criteria: A Cross-Sectional Study of Lifestyle. J Periodontol. 2017 Jun;88(6):602-609. doi: 10.1902/jop.2017.160426. Epub 2017 Jan 27. PMID 28128681
- [Background] Hansen GM, Egeberg A, Holmstrup P, Hansen PR. Relation of Periodontitis to Risk of Cardiovascular and All-Cause Mortality (from a Danish Nationwide Cohort Study). Am J Cardiol. 2016 Aug 15;118(4):489-93. doi: 10.1016/j.amjcard.2016.05.036. Epub 2016 May 30. PMID 27372888
- [Background] Holmstrup P, Damgaard C, Olsen I, Klinge B, Flyvbjerg A, Nielsen CH, Hansen PR. Comorbidity of periodontal disease: two sides of the same coin? An introduction for the clinician. J Oral Microbiol. 2017 Jun 14;9(1):1332710. doi: 10.1080/20002297.2017.1332710. eCollection 2017. PMID 28748036
- [Background] Hansen PR, Holmstrup P. Cardiovascular Diseases and Periodontitis. Adv Exp Med Biol. 2022;1373:261-280. doi: 10.1007/978-3-030-96881-6_14. PMID 35612803
- [Background] Joseph R, Rajappan S, Nath SG, Paul BJ. Association between chronic periodontitis and rheumatoid arthritis: a hospital-based case-control study. Rheumatol Int. 2013 Jan;33(1):103-9. doi: 10.1007/s00296-011-2284-1. Epub 2012 Jan 7. PMID 22228465
- See also: Related Info — http://odont.ku.dk/fagomr/parodontologi/